CLINICAL TRIAL: NCT02957929
Title: A Phase 1, Randomized, Placebo-Controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Oral Doses of APX001, to Investigate the Effect of Food on APX001 and to Investigate the Drug-Drug Interaction Potential of APX001
Brief Title: Safety, Pharmacokinetics, Bioavailability, Food Effect, Drug-Drug Interaction Study of APX001 Administered Orally
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: APX001-102; C4791002 (Other: Alias Study Number)
Record Dates: First submitted 2016-11-01; First posted 2016-11-08 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Cohort 1a, Period A (Experimental): single intravenous dose, crossover
  Interventions: Drug: APX001 single IV dose; Drug: Matching placebo control
- Cohort 1a, Period B (Experimental): single oral dose, crossover
  Interventions: Drug: APX001 single oral dose 1; Drug: Matching placebo control
- Cohort 1a, Period C (Experimental): single oral dose
  Interventions: Drug: APX001 single oral dose 2; Drug: Matching placebo control
- Cohort 1a, Period D (Experimental): single oral dose, crossover
  Interventions: Drug: APX001 single oral dose 3; Drug: Matching placebo control
- Cohort 1b, Period E (Experimental): Single oral dose under fasted conditions, crossover
  Interventions: Drug: APX001 single oral dose fasted; Drug: Matching placebo control
- Cohort 1b, Period F (Experimental): Single oral dose under fed conditions, crossover
  Interventions: Drug: APX001 single oral dose fed; Drug: Matching placebo control
- Cohort 2 (Experimental): Multiple oral doses
  Interventions: Drug: APX001 multiple oral doses 1; Drug: Matching placebo control
- Cohort 3 (Experimental): Multiple oral doses
  Interventions: Drug: APX001 multiple oral doses 2; Drug: Matching placebo control
- Cohort 4 (Experimental): Multiple oral doses in presence of CYP probe substrates
  Interventions: Drug: APX001 single IV dose; Drug: APX001 multiple oral doses 3; Drug: Cytochrome P450 substrates

INTERVENTIONS:
Drug: APX001 single IV dose
  Arms: Cohort 1a, Period A; Cohort 4
Drug: APX001 single oral dose 1
  Arms: Cohort 1a, Period B
Drug: APX001 single oral dose 2
  Arms: Cohort 1a, Period C
Drug: APX001 single oral dose 3
  Arms: Cohort 1a, Period D
Drug: APX001 single oral dose fasted
  Arms: Cohort 1b, Period E
Drug: APX001 single oral dose fed
  Arms: Cohort 1b, Period F
Drug: APX001 multiple oral doses 1
  Arms: Cohort 2
Drug: APX001 multiple oral doses 2
  Arms: Cohort 3
Drug: APX001 multiple oral doses 3
  Arms: Cohort 4
Drug: Cytochrome P450 substrates
  Arms: Cohort 4
Drug: Matching placebo control
  Arms: Cohort 1a, Period A; Cohort 1a, Period B; Cohort 1a, Period C; Cohort 1a, Period D; Cohort 1b, Period E; Cohort 1b, Period F; Cohort 2; Cohort 3

SUMMARY:
This is a Phase l double-blind, placebo-controlled, randomized study to investigate the safety, tolerability, pharmacokinetics, bioavailability and food effect of single doses of APX001 administered intravenously and orally, followed by an evaluation of the safety, tolerability, pharmacokinetics and drug-drug interaction potential of multiple doses of APX001 administered orally.

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing potential must agree to avoid pregnancy during the study and to use contraception at least 2 weeks before the start of the study until 3 months after the last dose of study drug.
* Males with partner(s) of childbearing potential must agree to use appropriate barrier contraception from the screening period until 3 months after the last dose of study drug.
* Screening hematology, clinical chemistry, coagulation and urinalysis consistent with overall good health.
* No significantly abnormal findings on physical examination, ECG and vital signs.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Any uncontrolled or active major systemic disease including, but not limited to: cardiovascular, pulmonary, gastrointestinal, metabolic, urogenital, neurological, immunological, psychiatric, or neoplastic disorder with metastatic potential.
* History or presence of malignancy within the past year. Subjects who have been successfully treated with no recurrence of basal cell carcinoma of the skin or carcinoma in-situ of the cervix may be enrolled.
* Use of prescription medication within 14 days prior to the first dose of study drug and throughout the study.
* Use of non-prescription or over-the-counter medications within 7 days prior to the first dose of study drug and throughout the study.
* Positive results on any of the following Screening laboratory tests: serum pregnancy test, urine alcohol test, urine drugs of abuse, hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single and multiple oral doses of APX001 as measured by adverse events (AEs), physical examinations (PE), vital signs (VS), laboratory safety tests, urinalysis and 12-lead electrocardiograms (ECG). | 21 days

SECONDARY OUTCOMES:
Pharmacokinetics of single and multiple doses of APX001 as measured by maximum observed concentration (Cmax). | 21 days
Pharmacokinetics of single and multiple dose of APX001 as measured by area under the curve (AUC). | 21 days
Pharmacokinetics of single and multiple doses of APX001 as measured by terminal half life (t1/2). | 21 days
Pharmacokinetics of single and multiple doses of APX001 as measured by volume of distribution (Vd). | 21 days
Pharmacokinetics of single and multiple doses of APX001 as measured by elimination rate constant (Kel). | 21 days
Pharmacokinetics of single and multiple doses of APX001 as measured by accumulation ratio. | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Marc Engelhardt, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (2):
- Netherlands (2):
  - PRA Health Sciences (PRA) - Early Development Services (EDS), Groningen
  - PRA Health Sciences, Groningen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hodges MR, Ople E, Wedel P, Shaw KJ, Jakate A, Kramer WG, Marle SV, van Hoogdalem EJ, Tawadrous M. Safety and Pharmacokinetics of Intravenous and Oral Fosmanogepix, a First-in-Class Antifungal Agent, in Healthy Volunteers. Antimicrob Agents Chemother. 2023 Apr 18;67(4):e0162322. doi: 10.1128/aac.01623-22. Epub 2023 Mar 29. PMID 36988461